CLINICAL TRIAL: NCT07255157
Title: Deciphering the Role of Peripheral Helper T-cells in Common Variable ImmunoDeficiency Pathophysiology in Patients With Non-infectious Complications
Brief Title: Peripheral Helper T-cells in Common Variable ImmunoDeficiency
Acronym: TAPDI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2025/037
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Common Variable Immunodeficiency
Keywords: common variable immunodeficiency; peripheral helper T cells; B cells
MeSH Terms: conditions — Common Variable Immunodeficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common variable immunodeficiency (Experimental)
  Interventions: Other: blood sample
- Controls (Active Comparator): Healthy controls
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — 48 ml whole blood for Peripheral blood mononuclear cell (PBMC) and serum isolation

SUMMARY:
The aim is to determine whether whether Tph could support non-infectious complications through providing help to pathological B-cells.

DETAILED DESCRIPTION:
Common variable immunodeficiency (CVID), the most common symptomatic primary immunodeficiency in adults, can associate recurrent infections with severe non-infectious complications. Unfortunately, there is still no absolute biomarker predicting which CVID patient will develop non-infectious complications. Thus, novel biomarkers which could help refining CVID patient prognosis require further investigations. Moreover, the immune mechanisms driving non-infectious complications remain elusive. Therefore, further insight into CVID pathophysiology is needed to discover new treatments for CVID patients with non-infectious complications (CVIDc). The preliminary results show that CVIDc patients have an increase of circulating peripheral helper T-cells (Tph) , in comparison with patients with infectious manifestations only (CVIDi) and healthy individuals (HI). Recently described, Tph express CXCR3, help memory B-cells and are found in inflamed tissues in auto-immune diseases. They represent a major reservoir of auto-reactive T-cells, suggesting that Tph are key to drive auto-immune processes. Some authors hypothesized that Tph can help atypical memory B-cells (ABCs), a B-cell subset which is involved in auto-immune disease pathophysiology and which is also expanded in CVIDc patients. The investigators observed that CXCR3+ cells were increased in the spleen of CVIDc patients in comparison with non-CVID controls. These CXCR3+ cells could correspond to Tph supporting extra-follicular reaction and then B-cell tolerance loss. The hypothesis is that alterations in T-B cell collaboration leads to the amplification of Tph in CVID patients. Tph could support non-infectious complications in target tissues through providing help to pathological B-cells such as ABCs. Using peripheral blood from CVIDc/CVIDi patients and HI, the investigators will determine whether Tph support pathological B cell activation in CVIDc patients using T-B co-cultures. Patients will be included during their routine follow-up, for one day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age ≥ 18 years;
* Standard criteria will be applied to diagnose CVID, specifically requiring: 1) low serum IgG level <5 g/L, combined with low IgM- and/or IgA-isotype concentrations <0.4 g/L or <0.7 g/L, respectively; 2) poor antibody responses to immunization or infection; and 3) exclusion of other defined forms of secondary hypogammaglobulinemias. Patients meeting the definitional criteria for CVID will be included, regardless of the duration of the disease or the treatment received (gammaglobulins substitution or not);
* Being affiliated to health insurance;
* Willing to participate and to sign informed consent.

Exclusion Criteria:

* Patients on corticosteroids and/or immunosuppressants;
* Patients with a primary immunodeficiency genetically characterized, such as Bruton disease our HyperIgM syndrome;
* Patients with an active chronic infection;
* Pregnant or breastfeeding women;
* Persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Ability of Tph to promote differentiation and antibody production by memory B cells (B-T co-culture) | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François VIALLARD, Prof, Principal Investigator — University Hospital, Bordeaux; Jonathan VISENTIN, Prof, Study Director — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de médecine interne, Pessac, France

IPD SHARING:
Plan to Share IPD: No